CLINICAL TRIAL: NCT01427673
Title: Phase III Single-blind Randomized Controlled Trial of Bipap Versus CPAP in Overlap Syndrome
Brief Title: Continuous Positive Airway Pressure Versus Noninvasive Ventilation in Patients With Overlap Syndrome
Acronym: OS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: United States Air Force (U.S. Federal Agency)
Collaborators: Landstuhl Regional Medical Center (U.S. Federal Agency); Good Samaritan Hospital (Unknown); Dayton Respiratory Center (Other); Tripler Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patrick F. Allan, Chief, Pulmonary, Critical Care and Sleep Medicine, United States Air Force
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USAF
Record Dates: First submitted 2011-08-29; First posted 2011-09-01 (Estimated); Last update posted 2011-09-01 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Obstructive Sleep Apnea; Overlap Syndrome
Keywords: Chronic Obstructive Pulmonary Disease; Obstructive Sleep Apnea; Overlap Syndrome; COPD; OSA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP Procedure control group (Active Comparator): Overlap patients randomly assigned to the CPAP titrated per AASM guidelines.
  Interventions: Procedure: Bipap procedure
- Bipap procedure group (Experimental): Overlap patients randomized to Bipap titrated per AASM guidleines with an IPAP to EPAP diffrence of at least 8 cm H2O.
  Interventions: Procedure: Bipap procedure

INTERVENTIONS:
Procedure: Bipap procedure — Overlap patients randomized to Bipap titrated per AASM guidleines with an IPAP to EPAP diffrence of at least 8 cm H2O.

SUMMARY:
The purpose of this study is to determine if Bipap should assume a standard-of-care role in the management of overlap syndrome.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a leading cause of disability and death worldwide. Acute exacerbations of COPD (AECOPD), in particular, serve as marker of an accelerated disease course and thus herald an increased risk of not only repetitive AECOPD episodes but also deteriorating pulmonary function and death (2). Obstructive sleep apnea (OSA), when it occurs in combination with COPD, is an increasingly recognized contributor to AECOPD episodes. OSA consists of repetitive sleep-related partial loss of airway caliber arising from increased transmural pressures which favor luminal collapse. OSA is estimated to afflict 4 to 9% of the populations, a prevalence which is anticipated to climb hand-in-hand with the rising incidence of obesity.

The combination of the two disorders, which has been arbitrarily labeled as Overlap Syndrome (OS), has been linked with greater elevations in arterial carbon dioxide tensions and pulmonary vascular resistance and lower arterial oxygen tensions than is seen with either of its component disorders in isolation. Elevated pulmonary artery pressures may progress to cause cor pulmonale, a process whereby compensatory right ventricle remodeling, hypertrophy, and eventually, florid heart failure. In the setting of OSA, the therapeutic gold standard is nightly continuous positive airway pressure (CPAP). Essentially, CPAP machines function by administering a single continuous positive pressure airflow to the person's airway via an appropriately fitted nasal mask. The applied pressure stents open partially occluded airway segments during sleep. Though effective in OSA and OS, it is increasingly realized that for OS patients there may exist a reduction not only in airway patency but also in ventilatory drive when sleeping such that means to augment per breath volumes may attain incremental benefits to the use of CPAP alone. Although CPAP is ineffective in COPD, Bipap has shown benefit suggesting that patient with OSA and COPD may derive an improvement in health-related outcomes by using a ventilation modality which addresses both of the underlying conditions.

Bipap functions by combining the single flow in CPAP with a second inspiratory pressure assist which not only overcomes sleep-related airway resistance but also increases the magnitude of each breath resulting in lower diurnal carbon dioxide tensions and pulmonary artery pressures. Bipap may harbor a mortality benefit in COPD; but the study results are conflicting. It is unclear if Bipap is more effective at treating OSA than usual CPAP. However, it is in the setting of OS that Bipap may assume a prominent role through its ability to address both disorders; CPAP for the OSA portion and an inspiratory pressure assist to ameliorate the COPD piece. Thus far no study has been conducted to address whether OS may derive a particular benefit from Bipap or, more specifically, examine whether Bipap may diminish the risk of AECOPD, or heart failure-related hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 35 years, the diagnosis of both OSA and COPD. OSA must have been diagnosed using an American Academy of Sleep Medicine (AASM)-protocol overnight Type I polysomnogram assessment with a resultant RDI of >5 events/hour in association with OSA-attributable diurnal symptoms.
* COPD must be diagnosed using American Thoracic Society (ATS)-protocol pulmonary function testing.
* Patients must have Global Obstructive Lung Disease (GOLD) stage II COPD FEV1/FVC < 70% predicted in conjunction with an FEV1 <80% predicted.
* The patient must have a > 10 pack years smoking history and a documented history of at least one exacerbation leading to treatment with systemic glucocorticoids or antibiotics or hospitalization within the previous year.

Exclusion Criteria:

* Significant diseases other than COPD, i.e. disease or condition which, in the opinion of the investigator, may have put the patient at risk because of participation in the study or may have influenced either the results of the study or the patients' ability to participate in the study
* Patients with a diagnosis of asthma
* Patients with a life-threatening pulmonary obstruction, or a history of cystic fibrosis
* Patients with known active tuberculosis
* Patients with brittle/unstable diabetes mellitus
* Patients with a history of and/or active significant alcohol or drug abuse. See exclusion criterion 1
* Patients with a history of myocardial infarction within the year prior to Visit 1
* Patients with cardiac arrhythmia that required medical or surgical treatment in the 3 months prior to enrollment
* Patients who had taken an investigational drug within 30 days or 6 half-lives (whichever is greater) prior to Visit 1
* Use of systemic corticosteroid medication at unstable doses (i.e., less than 6 weeks on stable dose) or at doses in excess of the equivalent of 10 mg prednisolone per day or 20 mg every other day
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e., oral contraceptives).
* Patients with any respiratory infection or COPD exacerbation in the 4 weeks prior to Visit 1 or during the run-in period should have been postponed. In the case of a respiratory infection or COPD exacerbation during the run-in period, the run-in period could have been extended up to 4 weeks
* Patients who, during their CPAP titration study are found to require such excessive CPAP pressures as to mandate a Bipap titration
* Patients with either Cheyne-stokes respiration noted on PSG assessment or a central sleep apnea with an associated central event index > 5 events/hour (using AASM central apnea/hypopnea scoring criteria)

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
The co-primary AECOPD and heart failure (AHF) outcome will be subdivided (see below). | 12 month intervention period
  Number of patients with events:
  Occurrence of at least 1 COPD exacerbation; Occurrence of at least 1 COPD exacerbation leading to hospitalization; Occurrence of premature discontinuation of CPAP or Bipap; Occurrence of at least one clinician-diagnosed acute or acute-on-chronic heart failure event; Occurrence of arrythmogenic events requiring either the outpatient initiation of a new non-B blocker antiarrythmic agent or hospitalization to treat an arrythmia;
  Number of events (stratified by number of events over the 12 month period)will also be measured.

SECONDARY OUTCOMES:
Difference in exertional and questionnaire-based quality-of-life indicators | 12 month intervention period
  Difference from baseline in 6 minute walk test distance, oxygen walk test-assessed supplemental oxygen requirements, St. George's Respiratory Questionnaire (SGRQ) and UCSD Shortness of breath questionnaire scores.
  Mortality (subdivided into the following) Cancer, No. CVS, No. Pulmonary, No. Other, No. All causes, No.
  Mean and median nightly number of hours used for each NIV modality
Safety outcome measures | 12 month intervention period
  * Serious adverse events
  * Adverse events leading to treatment discontinuation
  * Treatment-related adverse events
  * Major adverse cardiovascular events (MACE) during treatment*
  * All-cause mortality with onset of fatal AECOPD during treatment with study intervention + 30 days *Included fatal cardiac disorders, fatal vascular disorders, sudden death, cardiac death, sudden cardiac death, serious adverse events (fatal and non-fatal) from myocardial infarction, and stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Wright-Patterson Medical Center, Wpafb, Ohio, United States

REFERENCES:
- [Result] Lee R. McNicholas WT. Obstructive sleep apnea in chronic obstructive pulmonary disease patients. Current Opinion in Pulmonary Medicine. 17(2):79-83, 2011. Hiestand D. Phillips B. The overlap syndrome: chronic obstructive pulmonary disease and obstructive sleep apnea. Critical Care Clinics. 24(3):551-63, vii, 2008. Owens RL. Malhotra A. Sleep-disordered breathing and COPD: the overlap syndrome. Respiratory Care. 55(10):1333-44; discussion 1344-6, 2010. Marin JM. Soriano JB. Carrizo SJ. Boldova A. Celli BR. Outcomes in Patients with Chronic Obstructive Pulmonary Disease and Obstructive Sleep Apnea The Overlap Syndrome. Am J Respir Crit Care Med Vol 182. pp 325-331, 2010.